CLINICAL TRIAL: NCT04987957
Title: Effect Of Musıc Therapy On Anxıety Levels In Prımary Care Famıly Health Workers In COVID-19 Pandemıc
Brief Title: Effect Of Musıc Therapy On Anxıety Levels In COVID-19 Pandemıc
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Saadet Can Çiçek, Assistant Proffessor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AIBU-SBF-SK-01
Record Dates: First submitted 2021-07-30; First posted 2021-08-03 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Anxiety
Keywords: Music Therapy
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: The sample groups of the research will be divided into two groups as experiment and intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): 4 music genres with expert opinion will be presented to the preference of the participants in the intervention group, these types of music; Classical Music, Turkish Classical Music, Turkish Folk Music and Sufi Music. The music is instrumental, 70 decibels and non-verbal. Participants will listen to a genre they choose and download to their mobile phones once for 5 days for 15 minutes. They will listen to the music in the environment they live in, at a time convenient for them, at the desired volume level and with headphones in accordance with the determined therapy program.
  At the beginning of the research, an Introductory Questionnaire will be applied to all participants. Trait Anxiety Inventory will be administered before music therapy on the 1st day of the study and after the music therapy application on the 5th day.
  Interventions: Other: Music Therapy
- Control group (No Intervention): No application will be made to the participants in the control group, and the data collection tools will be applied with the same frequency as in the intervention group.

INTERVENTIONS:
Other: Music Therapy — Classical Music, Turkish Classical Music, Turkish Folk Music and Sufi Music
  Arms: Experimental group

SUMMARY:
This study, which has a randomized controlled experimental design, was planned to determine the effect of music therapy on the anxiety level of family health personnel working in primary health care centers during the COVID-19 pandemic. The study will be carried out between 4 August and 31 December with nurses, midwives and other family health personnel working in family health centers. Participants will be randomized into two groups, a control and an intervention group. Individuals in the intervention group will receive 15 minutes of music therapy once a day for 5 days. No intervention will be made in the control group. Data Descriptive Question and State-Trait Anxiety Inventory online design; It will be collected on the Google Forms platform.. Data analysis will be done using SPSS 20 program.

DETAILED DESCRIPTION:
Today, billions of people are struggling with the pandemic caused by the COVID-19 virus. The pandemic causes many psychosocial and mental health problems in humans. (Montano and Acebes 2020, Guo, Feng et al. 2020, Ostacoli, Cosmo et al. 2020, Carmassi, Foghi et al. 2020, Heitzman 2020, Sun, Sun et al. 2021, Yuan ,Gong et al. 2021, Taylor, Landry et al 2020 ). Many people have faced problems such as stress, depression and anxiety (Liu, Yang et al 2020). Compared to other segments of the society, health workers experience these problems more frequently and more severely. The reason for this is that healthcare professionals undertake the task of providing health care services to people infected with the virus, being together with patients, having close contact and meeting their health needs. This situation triggers the risk of contact with patients, fear of death, concerns about the health of themselves and their family members, and psychological problems (Aykurt and Aykurt 2020). Therefore, healthcare workers are considered to be a high-risk group in which the psychological consequences of COVID-19 are significant and persistent (Fiorillo and Gorwood 2020).

Studies in the literature have shown that healthcare workers experience severe anxiety due to COVID-19. (Yanez, Jahanshahi et al 2020, Sahebi, Nejati et al 2021, Lai, Ma et al 2019, Ataç, Sezerol et al 2020, Luo, Liu et al 2021).

It is very important to screen health workers who provide uninterrupted service in pandemic conditions in terms of anxiety and other psychological problems and to plan remedial interventions. In this context, music therapy, which is known as an effective method to reduce the anxiety level of individuals and reduce stress, comes to mind. Music therapy studies with healthcare professionals are limited in the literature. In this context, it is aimed that this study will contribute to filling this gap in the literature and creating a database.

ELIGIBILITY:
Inclusion Criteria:

* Not having a verbal or auditory communication barrier,
* To voluntarily agree to participate in the research,
* Not having a diagnosis of neuropsychiatric disease,
* Having the opportunity to fill out the surveys online,
* Possess the title of midwife or nurse.

Exclusion Criteria:

* Having a diagnosed neuropsychiatric disorder,
* Verbal and auditory communication disability,
* Not being willing to participate in the research,
* Having a title other than a midwife or nurse.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2021-12-08 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Two months
  State-Trait Anxiety Scale
  The scale consists of a total of 40 items in two separate parts. The scale includes direct and reversed statements. The total score that can be obtained from the scale is a minimum of 20 and a maximum of 80 points, and an increase in the score indicates an increase in the level of anxiety (Öner and Le Compte 1983).

CONTACTS AND LOCATIONS:
Overall Officials: Saadet Can Çiçek, Study Director — http://www.ibu.edu.tr/tr
Locations (1):
- Family Health Centers in Bolu, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No